CLINICAL TRIAL: NCT00005778
Title: Randomized Trial of High-Dose IV Cyclophosphamide Versus Monthly IV Cyclophosphamide
Brief Title: High-Dose Intravenous (IV) Cyclophosphamide Versus Monthly IV Cyclophosphamide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Michelle Petri Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: N01 AR92243; NIAMS-046
Record Dates: First submitted 2000-06-03; First posted 2000-06-05 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Systemic Lupus Erythematosus (SLE); Cytoxan; Cyclophosphamide; High-dose immunoablative therapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic

INTERVENTIONS:
Drug: High-dose immunoablative therapy — 1. High dose cyclophosphamide for 4 days.
  2. NIH monthly IV cytoxan for 6 months followed by quarterly for 2 years.

SUMMARY:
This study compares the effectiveness of high-dose cyclophosphamide treatment with the "gold standard" treatment, monthly intravenous (IV) cyclophosphamide, in people with moderate to severe lupus that does not respond to high-dose corticosteroid therapy. We will give patients either IV cyclophosphamide (750 milligrams per square meter of body surface area) monthly for 6 months, followed by quarterly maintenance therapy, or high-dose IV cyclophosphamide (50 milligrams per kilogram body weight per day) for the first four days of the study. Patients will be followed for 24 months after therapy.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE or lupus) remains the prototypic autoimmune disease. Recent data show that its incidence has tripled since 1970 and its prevalence is 1 in 800 in Rochester, Minnesota. The natural history of lupus in our cohort is one of (1) relapsing/ remitting or (2) chronic activity, with only 17 percent of patients having periods of long quiescence. Over 75 percent of our African-American patients and 50 percent of our Caucasian patients have renal (kidney) involvement. Over 50 percent suffer permanent damage in one or more organ systems, and over 15 percent have renal failure.

Researchers at the National Institutes of Health (NIH) have shown that, for patients with severe lupus, especially with renal involvement, monthly IV pulse cyclophosphamide (500 to 1000 mg/m squared BSA) for 6 months followed by quarterly maintenance for 2 years is superior to high-dose corticosteroid treatment. NIH and others have shown that IV pulse cyclophosphamide is also effective for severe lupus in other organs. However, even monthly IV cyclophosphamide is not successful in all cases, and it, too, has associated toxicity, especially premature ovarian failure. For that reason, we have pioneered the use of high-dose immunoablative cyclophosphamide (200 mg/kg) in 10 patients with severe lupus refractory to other treatments.

Because of the initial success of this approach, including 75 percent complete response (on no medications) in renal lupus, we are conducting a controlled trial of high-dose immunoablative cyclophosphamide versus the "gold standard" monthly IV cyclophosphamide in people with moderate to severe lupus refractory to high-dose corticosteroid therapy. We will give patients either 750 mg/m2 of body surface area IV cyclophosphamide monthly for 6 months, followed by quarterly maintenance therapy (we will readmit patients, if necessary, for infections or other complications) or cyclophosphamide 50 mg/kg/d intravenously on days 1-4. We will calculate the dose of cyclophosphamide according to ideal body weight. Patients are scheduled to receive only one course of therapy. We will follow patients according to the infective guidelines for BMT.

ELIGIBILITY:
All patients with moderate-to-severe SLE will be considered for this trial, including women and minorities. SLE is too rare a disease in children for it to be feasible to include them. Patients must meet the following criteria to be eligible for participation in this clinical trial:

* Four or more ACR criteria (90), as revised by Hochberg (91) for the classification of SLE.
* Involvement of one or more of the following organ systems (renal, neurologic, hematologic, cardiac, pulmonary, cutaneous, gastrointestinal) of moderate-to-severe severity as indicated by an "A" score on the BILAG, a "2" or "3" for severity on SLAM, or severe enough to require hospitalization if the organ involvement was not "captured" on either the BILAG or SLAM instruments.
* A lack of response to daily corticosteroids in moderate-to-high doses (0.5 -1 mg prednisone/kg/day or equivalent anti-inflammatory dose of methyprednisolone, dexamethasone, or triamicinolone). When cyclophosphamide is the accepted standard of care (renal and neurologic), the maximally tolerated dose of prednisone will be sufficient to meet the corticosteroid criterion. The ideal body weight will be used for this criterion in patients who are morbidly obese. The equivalent dose of triamcinolone (4mg triamcinolone=5mg prednisone) can be used to meet the criterion.

And/or:

* A lack of response to IV pulse corticosteroids (1 gram methylprednisolone or 180 mg dexamethasone).
* Duration of treatment to determine lack of response is 3 days or longer for neurologic, renal, hematologic, pulmonary, or cardiac lupus, one month or longer for serositis.

And/or:

* Equivalent degree of immunosuppression with azathioprine, methotrexate, cyclosporin, or mycophenolate mofetil. Equivalent degrees of immunosuppression are: azathioprine - 100 mg daily or more; methotrexate - 7.5 mg weekly or more; cyclosporin - 150 mg daily or more; mycophenolate mofetil - 1000 mg daily or more. Duration to determine lack of response should be one month or longer.

And/or:

* Appropriate other treatment (such as intravenous immunoglobulin for hemolytic anemia and thrombocytopenia).
* SLE patients seeking treatment for neurological complaints will be evaluated by a neurologist to concur that the patient meets eligibility criteria.
* Appropriate other treatment for cutaneous lupus patients may include combination antimalarial drugs (such as the combination of hydroxychloroquine or chloroquine with quinacrine).
* Patients may enter the trial if they received one dose of IV cyclophosphamide to "temporize" or "stablize" them prior to screening visit or after signing consent or if previous IV cyclophosphamide was for a PAST organ system, and patient presents with NEW organ system requiring IV cyclophosphamide.
* Insurance or other source of funds to pay for expenses related to this trial.

Exlcusion Criteria:

* Age less than 18 years and over 70 years.
* Any risk of pregnancy - ALL female patients must have an effective means of birth control or be infertile due to hysterectomy, fallopian tube surgery, or menopause.
* Previous completion of the NIH IV cyclophosphamide protocol.
* Cardiac ejection fraction < 45%.
* Serum creatinine > 3.0 mg/dL.
* FVC or FEV < 50% predicted.
* Bilirubin > 2.0, transaminases > 2x normal.
* Patients who are preterminal or moribund.
* SLE patients presenting with arthritis for entry organ system.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2000-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
RIFLE | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Petri, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins University Division of Rheumatology, Baltimore, Maryland
  - Drexel University School of Medicine, Division of Hematology/Oncology, Philadelphia, Pennsylvania
  - Medical College of Wisconsin, Division of Rheumatology, Milwaukee, Wisconsin

REFERENCES:
- [Background] Brodsky RA, Petri M, Smith BD, Seifter EJ, Spivak JL, Styler M, Dang CV, Brodsky I, Jones RJ. Immunoablative high-dose cyclophosphamide without stem-cell rescue for refractory, severe autoimmune disease. Ann Intern Med. 1998 Dec 15;129(12):1031-5. doi: 10.7326/0003-4819-129-12-199812150-00007. PMID 9867758
- [Background] Brodsky RA, Sensenbrenner LL, Jones RJ. Complete remission in severe aplastic anemia after high-dose cyclophosphamide without bone marrow transplantation. Blood. 1996 Jan 15;87(2):491-4. PMID 8555470
- [Background] Brodsky RA, Smith BD. Bone marrow transplantation for autoimmune diseases. Curr Opin Oncol. 1999 Mar;11(2):83-6. doi: 10.1097/00001622-199903000-00002. PMID 10188071
- [Background] Levite M, Zinger H, Zisman E, Reisner Y, Mozes E. Beneficial effects of bone marrow transplantation on the serological manifestations and kidney pathology of experimental systemic lupus erythematosus. Cell Immunol. 1995 Apr 15;162(1):138-45. doi: 10.1006/cimm.1995.1061. PMID 7704902
- [Background] Petri M, Jones RJ, Brodsky RA. High-dose cyclophosphamide without stem cell transplantation in systemic lupus erythematosus. Arthritis Rheum. 2003 Jan;48(1):166-73. doi: 10.1002/art.10752. PMID 12528116
- [Background] Petri M. Cyclophosphamide: new approaches for systemic lupus erythematosus. Lupus. 2004;13(5):366-71. doi: 10.1191/0961203303lu1028oa. PMID 15230294